CLINICAL TRIAL: NCT02938988
Title: Full-mouth Antimicrobial Photodynamic Therapy as an Adjunct to Non-surgical Periodontal Disease Treatment in Down's Syndrome Patients
Brief Title: Antimicrobial Photodynamic Therapy as an Adjunct Treatment for Periodontal Disease in Down's Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOBDownSyndrome
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Periodontal Diseases
Keywords: Periodontal Diseases; Down Syndrome
MeSH Terms: conditions — Periodontal Diseases; Down Syndrome | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): Scaling and root planning and antimicrobial photodynamic therapy with red laser (658nm; 0.1W; 2229J/cm², 10s per point) and methylene blue dye (100μg/ml). Repetition after 3, 7 and 14 days.
  Interventions: Procedure: Antimicrobial photodynamic therapy; Procedure: Scaling and root planning; Device: red laser; Drug: methylene blue dye
- Control Group (Active Comparator): Scaling and root planning Repetition after 3, 7 and 14 days.
  Interventions: Procedure: Scaling and root planning

INTERVENTIONS:
Procedure: Antimicrobial photodynamic therapy — Described in arm/group
  Arms: Test group
Procedure: Scaling and root planning — Described in arm/group
Device: red laser — 658nm; 0.1W; 2229J/cm², 10s per point
  Arms: Test group
Drug: methylene blue dye
  Arms: Test group

SUMMARY:
The aim of this study was to evaluate the effectiveness of antimicrobial photodynamic therapy as an adjuvant of scaling and root planning for treatment of periodontal disease in patients with Down's Syndrome. After scaling and root planning, half of patients received antimicrobial photodynamic therapy with methylene blue dye and laser and the sessions were repeated after 3, 7 and 14 days. The other half received only scaling and root planning.

.

DETAILED DESCRIPTION:
Antimicrobial photodynamic therapy (aPDT) has been widely used in Periodontics to obtain reduction of periodontopathogenic bacteria with absence of systemic side effects and minimal bacterial resistance. Therefore, a good adjuvant alternative for periodontal disease treatment arises, especially for patients with Down syndrome (DS) who present greater severity and high prevalence of periodontal disease. Usually aPDT is used as an adjunct therapy to scaling and root planning.

ELIGIBILITY:
Inclusion Criteria:

Down's Syndrome Diagnose characterized by the whole chromosomal aneuploidy 15 to 52 years Absence of severe hearing loss could impair the comprehension about the dental treatment Absence of severe visual loss that could impair the comprehension about the dental treatment Presence of at least four teeth being one for hemiarch. Diagnose of gingivitis and periodontitis Absence of acute periodontal disease and necrotizing periodontal disease

Exclusion Criteria:

Smokers Use of alcohol Menopause Pregnancy Absence of all teeth Uncontrolled diabetes mellitus Uncontrolled hyperthyroidism Angina Uncontrolled hypertension Coagulopathy Use of illicit drugs Head and neck radiotherapy Chemotherapy Non-cooperative patients or patients with other diseases as autism.

Ages: 15 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Periodontal disease (gingivitis and periodontitis) measured by a periodontal probe and classified according to severity | one year
  Severe periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with clinical attachment level (CAL) ≥ 6mm and ≥1 interproximal site with periodontal probing depth (PPD) ≥5mm. Moderate periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with CAL ≥ 4mm or ≥ 2 interproximal sites in different teeth with PPD ≥5mm. Mild periodontitis was defined as ≥ 2 interproximal sites in different teeth with ≥ 3 mm CAL and ≥ 2 interproximal sites in different teeth with ≥ 4 mm PPD or at least 1 site with PPD ≥ 5 mm (20,21). Gingivitis was determined as follows: Subjects were considered healthy if presented PPD ≤3mm/ Bleeding on probing (BOP) extent scores < 10% and with gingivitis if presented PPD ≤3mm/ BOP extent scores >10%. Prevalence of periodontal disease was the sum of gingivitis, mild, moderate and severe periodontitis.

SECONDARY OUTCOMES:
Obesity measured by a tape and a scale | one day
  Obese if: body mass index - BMI ≥ 25 Kg/m2 (weight in kilograms, height in meters) Obese if: waist-to-hip ratio - WHR >0.85 for women. >0.9 for men. (measurement in centimeters) Obese if: waist circumference - > 80 cm for women and >94 cm for men.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira R, Michel RC, Greghi SL, Resende ML, Sant'Ana AC, Damante CA, Zangrando MS. Prevention and Periodontal Treatment in Down Syndrome Patients: A Systematic Review. PLoS One. 2016 Jun 29;11(6):e0158339. doi: 10.1371/journal.pone.0158339. eCollection 2016. PMID 27355338
- [Background] Martins F, Simoes A, Oliveira M, Luiz AC, Gallottini M, Pannuti C. Efficacy of antimicrobial photodynamic therapy as an adjuvant in periodontal treatment in Down syndrome patients. Lasers Med Sci. 2016 Dec;31(9):1977-1981. doi: 10.1007/s10103-016-2020-x. Epub 2016 Jul 6. PMID 27384040